CLINICAL TRIAL: NCT07063160
Title: Effect of Acupressure Therapy on Pain, Injection Fear, and Post-Injection Satisfaction in Patients Undergoing Intramuscular Injection
Brief Title: Effect of Acupressure Therapy on Pain, Fear, and Post-Injection Satisfaction in Patients Undergoing IM Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Onur Soydinç, Msc, Eastern Mediterranean University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EasternMUonur
Record Dates: First submitted 2025-02-22; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Injection Fear; Injection Site
Keywords: Intramuscular injection; Acupressure therapy; Pain; Injection Fear; Satisfaction
MeSH Terms: conditions — Iatrophobia; Pain; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intramuscular injection after acupressure therapy (Experimental): Before the injection is applied to the patients in the experimental group; First, the patient who filled in the Personal Information Form will first apply pressure with the thumb for 1 minute to the GB 30 point located at the junction between the medial two-thirds and the lateral one-third of a line connecting the greater trochanter and the sacral hiatus with the acupressure therapy method. Then, the Injection Fear Scale will be filled in. Then, Diclofenac Sodium injection will be applied IM. After the injection, the pain intensity will be measured with VAS and finally the Post-Injection Satisfaction Scale will be filled in.
  Interventions: Behavioral: Pain; Behavioral: Fear of injection; Behavioral: Post-injection satisfaction
- Intramuscular injection after standard application (Active Comparator): Before the injection to the patients in the control group; Personal Information Form and Injection Fear Scale will be filled. Then, Diclofenac Sodium injection will be applied IM without any therapy method. The patient whose pain intensity is measured with VAS after the injection will finally fill out the Injection Satisfaction Scale.
  Interventions: Behavioral: Pain; Behavioral: Fear of injection; Behavioral: Post-injection satisfaction

INTERVENTIONS:
Behavioral: Pain — Injection was used to determine the level of pain
Behavioral: Fear of injection — The scale developed determines the fear levels of individuals towards the injection procedure. The scale consists of 14 items. It was developed on a 5-point Likert type, 1-I am not afraid at all, 5- I am very afraid. The scale is calculated based on the item score average. The lowest score that can be obtained from the scale is 1, and the highest score is 5. As the score obtained from the scale increases, the level of fear increases. Stated in their research that the Cronbach Alpha value for the entire scale was 0.92.
Behavioral: Post-injection satisfaction — The scale developed to determine the satisfaction levels of patients regarding the injection process. The scale was developed in a 5-point Likert type, 1-I am not satisfied at all, 5-I am very satisfied. The scale is calculated based on the item score average. The lowest score that can be obtained from the scale is 1, and the highest score is 5. As the score obtained from the scale increases, the level of satisfaction increases. Post-injection satisfaction Scale consists of 9 items. In the study conducted, it was determined that the Cronbach Alpha value of the entire scale was 0.895.

SUMMARY:
The pain that develops when the needle is inserted into the muscle in an Intramuscular injection triggers anxiety in many people and can cause a lifelong fear of Intramuscular injection. Fear related to Intramuscular injection can result in postponing or not having the injection. Injection applications can also cause an increase in pain, fear and anxiety levels in individuals and a decrease in comfort and satisfaction levels. For this reason, nurses are expected to take precautions or implement interventions that will reduce pain, increase comfort and satisfaction, and alleviate the patient's symptoms during drug administration. The use of acupressure therapy can be effective in reducing the feeling of pain and alleviating/eliminating the fear felt against the injection and thus increasing satisfaction after the injection.

DETAILED DESCRIPTION:
Intramuscular (IM) injection is a parenteral drug application where large amounts of drugs are administered into the deep muscle layer. IM injections are frequently made into the Ventrogluteal (VG), Dorsogluteal (DG), Vastus Lateralis/LateroFemoral and Deltoid muscles. Studies conducted in recent years in particular have indicated that the DG region is a risky area due to its proximity to the gluteal artery and sciatic nerve, and therefore it is emphasized that it should not be preferred unless necessary. Although it is a frequently preferred application among drug administration methods, IM injections have serious risks such as "accidental administration of the drug into the vein and nerve damage, post-injection pain, ecchymosis, and swelling". One of the most common complications encountered in intramuscular injection applications is pain. Although pain is defined as a universal experience that every individual has encountered at least once in their life, there are individual differences in the perception and expression of pain. It is reported that the pain that occurs with IM injection is related to the mechanical trauma that occurs at the needle entry and the sudden pressure created by the drug while it is injected into the muscle. In IM injection applications, the patient's anxiety and fear level before the injection significantly affects the pain they feel. In IM injection applications, the pain that occurs when the needle is inserted into the muscle initiates anxiety and can also cause people to feel fear of IM injection applications throughout their lives. Due to the fear that develops due to IM injection, patients may postpone the injection application or do not have the injection. Injection applications may also cause an increase in pain, fear and anxiety levels and a decrease in comfort and satisfaction levels in individuals. For this reason, nurses are expected to take precautions or implement interventions that will reduce pain, increase comfort and satisfaction, and alleviate the patient's symptoms during drug applications. In the literature, there are applications such as using the appropriate injection technique, positioning the patient appropriately, slowly administering the drug to the tissue, using the Z technique, applying an air lock, diverting the patient's attention, and using different alternative therapy methods to reduce the pain that occurs due to injection applications. One of these alternative therapy methods is acupressure therapy.

Acupressure therapy is a technique that aims to relieve or prevent pain by applying pressure to certain points with fingers. The physiological effect of this method is associated with the stimulation of pain modulation through different mechanisms. It is accepted that the life energy called "Chi" flows along energy channels called "meridians" in the body, which are named according to the internal organs. There are 14 meridians in the human body, 12 of which are double and 2 are single. The pressure applied to the points on these channels reduces the tension in various parts of the body and the tension in the muscles, increases the secretion of endorphins and blood circulation. Acupressure application is based on applying manual pressure to the same point with the finger and palm for approximately 1 minute.

The American Pain Management Nursing Association has emphasized that correct and effective interventions should be applied to the patient, situation, environment and needs in order to manage pain/fear/anxiety and ensure patient satisfaction before, during and after interventional applications for patients. Before the intramuscular injection, most patients are afraid because they think they will feel pain, and they postpone or do not have the medication applied. This situation causes the treatment to be interrupted and the recovery to be delayed. At this point, the use of acupressure therapy can be effective in reducing the feeling of pain and alleviating/eliminating the fear felt against the injection and thus increasing the satisfaction after the injection. When the literature is examined, it is seen that the studies on the pain, fear of injection and the level of satisfaction after the injection in acupressure therapy in intramuscular injection applications are limited. In this context, this study was planned to examine the effect of acupressure therapy on pain, fear of injection and the level of satisfaction after the injection in patients who receive intramuscular injection.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be 18 years of age or older,

  * Have the physical and mental capacity to correctly evaluate the Visual Analog Scale (VAS),
  * Have the capacity to read and understand the research guidelines,
  * Have a prescription from the physician that only requests Diclofenac Sodium by Intra Muscular,
  * Have their treatment just started,
  * Be within the normal weight-obese range according to the BMI determined by the World Health Organization,
  * Have not received Intramuscular injections from the Ventrogluteal (VG) region in the last 6 months,
  * Have no scars, scar tissue, etc. in the VG region

Exclusion Criteria:

* - Using any painkillers on the day of the injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale pain scores of patients in the experimental group who received acupressure treatment after intramuscular injection | 1 day
  Visual Analog Scale score
Injection Fear Scale scores of patients in the experimental group who received acupressure treatment after intramuscular injection | 1 day
  Injection Fear Scale score
Post-Injection Satisfaction Scale scores of patients in the experimental group who received acupressure treatment after intramuscular injection | 1 day
  Satisfaction Scale scores

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Mediterranean University, Mersin, - Please Select -, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Yes

REFERENCES:
- [Result] Ayinde O, Hayward RS, Ross JDC. The effect of intramuscular injection technique on injection associated pain; a systematic review and meta-analysis. PLoS One. 2021 May 3;16(5):e0250883. doi: 10.1371/journal.pone.0250883. eCollection 2021. PMID 33939726
- [Result] Fu Q, Xie H, Zhou L, Li X, Liu Y, Liu M, Wang C, Wang X, Wang Z, Tang J, Xiao H, Xiao Z, Zhou J, Feng C, Wang L, Ao Z, Chen X, Su C, Wu X, Zhao M, Hu S, Lin H, Huang J, Xu G, Zhang Q, Jiang L. Traditional Chinese medicine auricular point acupressure for the relief of pain, fatigue, and gastrointestinal adverse reactions after the injection of novel coronavirus-19 vaccines: a structured summary of a study protocol for a multicentre, three-arm, single-blind, prospective randomized controlled trial. Trials. 2021 Feb 25;22(1):162. doi: 10.1186/s13063-021-05138-3. PMID 33632286
- [Result] Sanlialp Zeyrek A, Takmak S, Kurban NK, Arslan S. Systematic review and meta-analysis: Physical-procedural interventions used to reduce pain during intramuscular injections in adults. J Adv Nurs. 2019 Dec;75(12):3346-3361. doi: 10.1111/jan.14183. Epub 2019 Sep 13. PMID 31452229
- [Result] Suhrabi Z, Taghinejad H. Effect of acupressure (UB32) on pain intensity in intramuscular injections. Iran J Nurs Midwifery Res. 2014 Jan;19(1):24-7. PMID 24554956
- [Result] Cmc S, Lord H, Vargese SS, Kurian N, Cherian SA, Mathew E, Fernandez R. Effectiveness of physical stimulation for reducing injection pain in adults receiving intramuscular injections: a systematic review and meta-analysis. JBI Evid Synth. 2023 Feb 1;21(2):373-400. doi: 10.11124/JBIES-20-00590. PMID 36758552
- [Result] Inangil D, Inangil G. The effect of acupressure (GB30) on intramuscular injection pain and satisfaction: Single-blind, randomised controlled study. J Clin Nurs. 2020 Apr;29(7-8):1094-1101. doi: 10.1111/jocn.15172. Epub 2020 Jan 20. PMID 31891437